CLINICAL TRIAL: NCT02643706
Title: Relationship Between the Gene Polymorphism of Aldehyde Dehydrogenase 2 and Contrast Induced Nephropathy
Brief Title: Relationship Between ALDH2 and CIN
Acronym: REACTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: Qiluexcellentyouth
Record Dates: First submitted 2015-12-19; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Aldehyde dehydrogenase 2; contrast induced nephropathy; Gene polymorphism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 ml vein blood samples were collected from peripheral vein before coronary angiography or percutaneous coronary intervention.The blood is used to detecte the renal function , the genotype of aldehyde dehydrogenase 2 and aldehyde dehydrogenase activity. Another 5 ml vein blood samples were collected from peripheral vein to detecte the renal function 24-72 hours after the surgery. The samples would be centrifuged and saved in a -80℃ ultra-low temperature refrigerator.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CIN: CIN was defined as an absolute increase in serum creatinine concentration of at least 0.5 mg/dL (44.2umol/l) or a relative rise of at least 25% from baseline on the follow-up blood sample drawn 24 to 72 hours after the operation.
- Control: The enrolled patients without CIN.

SUMMARY:
The purpose of this clinical trial is to investigate the relationship between the gene polymorphism of aldehyde dehydrogenase 2 and contrast induced nephropathy and its mechanism.

DETAILED DESCRIPTION:
Patients undergoing coronary angiography or percutaneous coronary intervention will be recruited in this study after they sign the informed consent.5ml venous blood was extracted from the peripheral vein before the operation to detect the renal function, the genotype and enzyme activity of aldehyde dehydrogenase 2 ,and the levels of oxidative stress and inflammation.Another 5ml venous blood was extracted from the peripheral vein 24-72 hours after the operation to detect the renal function and the levels of oxidative stress and inflammation.Activated oxygen protein products , 4-HNE and hs-CRP as markers for oxidative stress and inflammation.The renal function index contains serum creatinine，urea nitrogen and cystatin C.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary intervention or coronary angiography at Yu Qilu hospital.
* All the patients or their guardians must sign the consent form before entering the trial.

Exclusion Criteria:

* Patients with acute renal failure, renal transplantation, end-stage renal disease, or dialysis treatment, GFR < 15ml/min.
* Use of renal toxicity drugs during the treatment, such as non steroidal anti-inflammatory drugs, etc.
* Patients who has used contrast agent 10 days before the operation.
* Cardiac shock, hypotension (systolic blood pressure < 95mmHg),or hyper- tension with difficulty to control.
* Allergy to contrast media.
* Congestive heart failure (left ventricular ejection fraction<40%), cardiac function NYHA grade IV.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective coronary intervention or coronary angiography in Qilu hospital from December 2015 to December 2016
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with different ALDH2 genotype | 1-30 days after samples collected
Change from baseline renal function after the operation | at admission and 24-72hours after coronary angiography or coronary intervention
  The baseline of renal function will be tested at the next morning after admission .The renal function will be tested again 24-72 hours after coronary angiography or coronary intervention.The changes of renal function will be recorded.The renal function index contains serum creatinine,urea nitrogen and cystatin C.

SECONDARY OUTCOMES:
Aldehyde dehydrogenase 2 activity | 1-30 days after samples collected
Activated oxygen protein products, 4-HNE and hs-CRP | 1-30 days after samples collected
  Activated oxygen protein products , 4-HNE and hs-CRP as markers for oxidative stress and inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Xu, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China